CLINICAL TRIAL: NCT03497312
Title: Assessment of Oral Health Related Quality of Life After Full Mouth Rehabilitation Under General Anesthesia in a Group of Egyptian Children With Special Health Care Need (A Before and After Study)
Brief Title: Assessment of Oral Health Related Quality of Life After Full Mouth Rehabilitation Under GA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Duha Mohammed abdelhameed, Doctor Duha Mohammed Abdelhameed pedodontist principle investigator, Cairo University
Other Study IDs: OHRQOL in SHCNC
Record Dates: First submitted 2018-04-02; First posted 2018-04-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Quality of Life
Keywords: Rehabilitation; children with disabilities; general anesthesia; Children with special healthcare need; handicapped children; full mouth rehabilitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: full mouth rehabilitation — full mouth rehabilitation under general anesthesia

SUMMARY:
To assess Oral health related quality of life (OHRQOL) after full mouth rehabilitation under GA in a group of Egyptian children with special healthcare need.

DETAILED DESCRIPTION:
* The study will be conducted in Department of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University, Egypt.
* Demographic variables (caregiver age and gender), socio-economic condition, , medical history, and dental history will be collected from the parent or caregiver. The height and weight of each child will be measured in the same manner to standardize the result and their body mass index will be calculated before and after in follow up period.
* On the day of the GA, parent or caregiver will complete questionnaires about their child's oral state and well-being over the previous 3 months and oral hygiene instructions will be given to the parent.
* The questionnaire will be delivered to the parents/caregivers at baseline and at the 6-month post-operative follow-up visit. Dental examination will be assessed at baseline (pre-operatively) and at 1,3, 6, months post-operative visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 5 to 14 years.
2. Diagnosed with physical, mental, or sensory disability (separately or combined).
3. Should have a minimum of 12 primary or permanent teeth, or a mixture that had not been treated within the past 12 months.

Exclusion Criteria:

1. Participation in any other concurrent clinical trials.
2. The presence of serious medical conditions or a transmissible disease such as malignant disease, hepatitis, AIDS etc.
3. Children whose parents had no home or mobile phone to enable post-operative contact.
4. Parent that will not sign the consent.

Ages: 5 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: Caregivers paired with their children with special health care needs attending Pediatric Dentistry and Dental Public Health department, faculty of dentistry, Cairo University Egypt, will be screened for diagnosis of their chief complaint. Patients will be enrolled in this study if they are compatible with eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2018-12-15 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Oral health related quality of life (OHRQOL) | at baseline and 6 month
  Oral health related quality of life (OHRQOL) will be measured by two validated questioner which are : Parental-Caregivers Perceptions Questionnaire (P-CPQ) and family impact scale(FIS). the unit of measurement is likert scale

SECONDARY OUTCOMES:
Body mass | at baseline and 6 month
  Body mass will be measure by body mass index,weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Sheriene Ezz Eldin, PHD, Study Director — Cairo University

REFERENCES:
- [Background] Baens-Ferrer C, Roseman MM, Dumas HM, Haley SM. Parental perceptions of oral health-related quality of life for children with special needs: impact of oral rehabilitation under general anesthesia. Pediatr Dent. 2005 Mar-Apr;27(2):137-42. PMID 15926291
- [Background] Gaynor WN, Thomson WM. Changes in young children's OHRQoL after dental treatment under general anaesthesia. Int J Paediatr Dent. 2012 Jul;22(4):258-64. doi: 10.1111/j.1365-263X.2011.01190.x. Epub 2011 Oct 17. PMID 21999137
- [Background] Jokovic A, Locker D, Stephens M, Kenny D, Tompson B, Guyatt G. Measuring parental perceptions of child oral health-related quality of life. J Public Health Dent. 2003 Spring;63(2):67-72. doi: 10.1111/j.1752-7325.2003.tb03477.x. PMID 12816135